CLINICAL TRIAL: NCT00761189
Title: An Open Label, Prospective, Non-comparative Study to Evaluate Flexible Dose of Paliperidone Extended-Release and Clinical Response in the Treatment of Subjects With Schizophrenia
Brief Title: PaliperidoNe Extended-Release [ER] Dosing and Clinical Response in Acute Schizophrenia
Acronym: PANDORA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015079; PAL-KOR-4001
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-01

CONDITIONS: Schizophrenia
Keywords: Paliperidone; R076477; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone (Experimental): Paliperidone extended-release (ER) tablet will be administered orally in dose range of 3 to 12 milligram (mg) per day for 12 weeks as per Investigator's discretion.
  Interventions: Drug: Paliperidone

INTERVENTIONS:
Drug: Paliperidone — Paliperidone extended-release (ER) tablet will be administered orally in dose range of 3 to 12 milligram (mg) per day for 12 weeks as per Investigator's discretion.
  Other Names: R076477; Invega extended-Release (ER) tablet

SUMMARY:
The purpose of this study is to evaluate the efficacy of paliperidone extended-release (ER) in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-centric (conducted in more than one center), prospective (study following participants forward in time), single arm, and non-comparative study of paliperidone Extended Release(ER) in participants with schizophrenia. The total study duration will be approximately of 104 weeks per participant. The study consists of following parts: Screening (that is, 14 days before study commences on Day 1); acute Treatment phase (single-oral dose of paliperidone for 12 weeks, dose ranging from 3 to 12 milligram); Extension phase 1 (12 weeks) and Maintenance treatment which will be followed by additional Extension phase 2 and long-term maintenance treatment. Efficacy of the participants will primarily be evaluated by Clinical Global Impression-Improvement (CGI-I) scale score. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Clinical Global Impression-Severity (CGI-S) score greater than or equal to 4 points (moderately ill) at Screening
* Childbearing potential women who consent to the consistent use of the acceptable contraception (oral contraceptive, contraceptive injection, intrauterine device, double barrier method and contraceptive patch)
* Participants who are capable of and willing to fill out the questionnaire for themselves
* Participants who are compliant with self-medication or can receive consistent help or support
* Have schizophrenia diagnosis by Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV)

Exclusion Criteria:

* Participants with the past history of neuroleptic malignant syndrome (NMS)
* Participants with Treatment Resistance history who have failed to be properly treated with more than two other kinds of antipsychotic agents (at least 4 weeks of the therapeutic dose administration)
* Participants with severe (pathologic or iatrogenic) gastrointestinal stenosis or participants who can not swallow the drug whole (The study drug must not be chewed, divided, melted or grinded because it can impact the study drug release profile.)
* Participants who have been exposed to the study drug within one month before screening
* Participants with significant risk including suicide or aggressive behavior

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (20):
- South Korea (20):
  - Bucheon-Si Gyeonggi-Do
  - Changnyung
  - Chunjoo
  - Daejeon
  - Daejun
  - Geonggi-Do
  - Gyeonggi-do
  - Incheon
  - Inchun
  - Jinju
  - Jungnam
  - Kwangjoo
  - Kyounggi
  - Kyunggi-Do
  - Kyungju
  - Kyungki
  - Kyunki
  - Pusan
  - Seoul
  - Ulsan

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone: Paliperidone extended-release (ER) tablet was administered orally in dose range of 3 to 12 milligram (mg) per day for 12 weeks as per Investigator's discretion.
Period: Overall Study
Arm/Group | Paliperidone
Started | 491
Completed | 306
Not Completed | 185
Not completed — Adverse Event | 42
Not completed — Lack of Efficacy | 45
Not completed — Lost to Follow-up | 36
Not completed — Withdrawal by Subject | 49
Not completed — Other | 13

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone
Number analyzed (Participants) | 491
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247
  Male | 244

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Assessed as Very Much Improved or Much Improved Based on Clinical Global Impression-Improvement (CGI-I) Scale - Intent-to-treat (ITT) Population
Description: The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: Week 12
Population: Intent to Treat (ITT) population for efficacy included all the eligible participants who received paliperidone extended-release (ER) at least once and who completed post baseline efficacy assessments.
Measure: Number; unit: Percentage of participants
Groups:
- Paliperidone Extended-release (ER): Paliperidone extended-release (ER) tablet was administered orally in dose range of 3 to 12 milligram (mg) per day for 12 weeks as per Investigator's discretion.
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 345
Percentage of participants | 34.78

2. Primary Outcome: Percentage of Participants Assessed as Very Much Improved or Much Improved Based on Clinical Global Impression-Improvement (CGI-I) Scale - Per Protocol (PP) Population
Description: as for outcome 1
Time Frame: Week 12
Population: Per protocol (PP) population included all the participants who received paliperidone extended-release (ER) at least once and who completed the clinical study without violating the study protocol.
Measure: Number; unit: Percentage of participants
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 260
Percentage of participants | 41.92

3. Secondary Outcome: Personal and Social Performance (PSP) Scale Score - Intent-to-treat (ITT) Population
Description: The PSP scale assesses the degree of dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (1, absent to 6, very severe) in each of the 4 domains. Participants with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; less or equal to 30, functioning so poorly as to require intensive supervision.
Time Frame: Baseline, Week 4 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 345
Units on a scale
  Baseline | 49.39 (14.69)
  Week 4 | 59.44 (13.54)
  Week 12 | 62.76 (13.93)

4. Secondary Outcome: Personal and Social Performance (PSP) Scale Score - Per Protocol (PP) Population
Description: as for outcome 3
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 260
Units on a scale
  Baseline | 49.70 (14.73)
  Week 4 | 60.27 (13.34)
  Week 12 | 64.73 (13.09)

5. Secondary Outcome: Percentage of Participants Continuously Treated With 6 Milligram Per Day Regimen Until Week 12 - Intent-to-treat (ITT) Population
Description: Percentage of participants who were continuously treated with paliperidone extended-release (ER) 6 milligram per day regimen until Week 12 are reported here.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 345
Percentage of participants | 38.84

6. Secondary Outcome: Percentage of Participants Continuously Treated With 6 Milligram Per Day Regimen Until Week 12 - Per Protocol (PP) Population
Description: as for outcome 5
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 260
Percentage of Participants | 41.54

7. Secondary Outcome: Drug Attitude Inventory (DAI) Score - Intent-to-treat (ITT) Population
Description: The DAI-10 is a 10-item questionnaire to assess 1) subjective experience of drug and 2) attitudes and beliefs toward neuroleptics which may influence compliance in schizophrenia participants. It is the binary scale assessing the participant's subjective response. A 'compliant' response is scored as +1; a dysphoric response is scored as -1. A positive sum of items indicates a positive subjective response (SR); a negative sum of scores indicates a negative SR (non-compliant). The final score is the grand total of the positive and negative points. Total score ranges from (-) 10 to (+) 10, higher score indicates positive SR (compliant) and lower score indicates negative SR (non-compliant).
Time Frame: Baseline, Week 4 and 12
Population: Intent to Treat (ITT) population for efficacy included all the eligible participants who received paliperidone extended-release (ER) at least once and who completed post baseline efficacy assessments. "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 343
Units on a scale
  Baseline | -2.34 (4.78)
  Week 4 | -3.37 (4.53)
  Week 12 | -3.57 (4.54)

8. Secondary Outcome: Drug Attitude Inventory (DAI) Score - Per Protocol (PP) Population
Description: as for outcome 7
Time Frame: Baseline, Week 4 and 12
Population: Per protocol (PP) population included all the participants who received paliperidone extended-release (ER) at least once and who completed the clinical study without violating the study protocol. "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 259
Units on a scale
  Baseline | -2.39 (4.81)
  Week 4 | -3.49 (4.53)
  Week 12 | -4.02 (4.26)

9. Secondary Outcome: Clinical Global Impression - Severity (CGI-S) Score - Intent-to-treat (ITT) Population
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 345
Units on a scale
  Baseline | 4.62 (0.70)
  Week 2 | 4.08 (0.81)
  Week 4 | 3.73 (0.87)
  Week 8 | 3.50 (0.91)
  Week 12 | 3.29 (0.98)

10. Secondary Outcome: Clinical Global Impression - Severity (CGI-S) Score - Per Protocol (PP) Population
Description: as for outcome 9
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 260
Units on a scale
  Baseline | 4.60 (0.68)
  Week 2 | 4.02 (0.81)
  Week 4 | 3.66 (0.85)
  Week 8 | 3.40 (0.87)
  Week 12 | 3.10 (0.91)

11. Secondary Outcome: Number of Participants With Categorical Scores Based on Clinical Global Impression - Improvement (CGI-I) Scale - Intent-to-treat (ITT) Population
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 345
Participants
  Very much improved | 5
  Much improved | 115
  Minimally Improved | 158
  No change | 46
  Minimally worse | 15
  Much worse | 6
  Very much worse | 0

12. Secondary Outcome: Number of Participants With Categorical Scores Based on Clinical Global Impression - Improvement (CGI-I) Scale - Per Protocol (PP) Population
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 260
Participants
  Very much improved | 5
  Much improved | 104
  Minimally Improved | 118
  No change | 28
  Minimally worse | 5
  Much worse | 0
  Very much worse | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Description: Safety population included all the eligible participants who received paliperidone extended-release (ER) at least once .
Arm/Group | Paliperidone
Serious Adverse Events (participants affected / at risk) | 55/491
Other Adverse Events (participants affected / at risk) | 243/491
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone (N=491)
Anaemia (Blood and lymphatic system disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest Discomfort (General disorders) | 1
Hepatic Steatosis (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1
Tendon Injury (Injury, poisoning and procedural complications) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Benign Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Dystonia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Tardive Dyskinesia (Nervous system disorders) | 1
Abnormal Behaviour (Psychiatric disorders) | 1
Acute Psychosis (Psychiatric disorders) | 1
Aggression (Psychiatric disorders) | 5
Agitation (Psychiatric disorders) | 1
Alcohol Abuse (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 4
Completed Suicide (Psychiatric disorders) | 1
Delusion (Psychiatric disorders) | 3
Hallucination (Psychiatric disorders) | 1
Hallucination, Auditory (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 1
Nicotine Dependence (Psychiatric disorders) | 1
Obsessive Thoughts (Psychiatric disorders) | 1
Obsessive-Compulsive Disorder (Psychiatric disorders) | 1
Psychotic Disorder (Psychiatric disorders) | 2
Schizophrenia (Psychiatric disorders) | 13
Schizophrenia, Paranoid Type (Psychiatric disorders) | 1
Social Avoidant Behaviour (Psychiatric disorders) | 3
Suicidal Ideation (Psychiatric disorders) | 1
Suicide Attempt (Psychiatric disorders) | 1
Treatment Noncompliance (Social circumstances) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone (N=491)
Constipation (Gastrointestinal disorders) | 46
Dry Mouth (Gastrointestinal disorders) | 49
Nasopharyngitis (Infections and infestations) | 10
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 30
Akathisia (Nervous system disorders) | 65
Dizziness (Nervous system disorders) | 13
Dizziness Postural (Nervous system disorders) | 24
Headache (Nervous system disorders) | 45
Sedation (Nervous system disorders) | 42
Somnolence (Nervous system disorders) | 42
Tremor (Nervous system disorders) | 35
Insomnia (Psychiatric disorders) | 97
Amenorrhoea (Reproductive system and breast disorders) | 21

LIMITATIONS AND CAVEATS:
Some Adverse Events summaries were reported based on estimates due to the fact that they were not prepared in the original study report and the relevant definitions of the data elements were not available for these summaries to be regenerated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less